CLINICAL TRIAL: NCT01827839
Title: Immunogenicity and Safety of GSK Biologicals' Herpes Zoster Vaccine GSK1437173A in Adults With a Prior Episode of Herpes Zoster
Brief Title: Immunogenicity and Safety of GlaxoSmithKline (GSK) Biologicals' Herpes Zoster Subunit (HZ/su) Vaccine GSK1437173A in Adults With a Prior Episode of Herpes Zoster
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 116796; 2012-003643-30 (EudraCT Number)
Record Dates: First submitted 2013-03-28; First posted 2013-04-10 (Estimated); Results first posted 2017-03-07 (Actual); Last update posted 2018-10-18 (Actual); Status verified 2017-10

CONDITIONS: Herpes Zoster
Keywords: Adults; Safety; Immunogenicity; Zoster
MeSH Terms: conditions — Herpes Zoster | interventions — Herpes Zoster Vaccine

ARMS (1):
- HZ Group (Experimental): Subjects will receive 2 doses of the HZ/su vaccine at Month 0 and Month 2.
  Interventions: Biological: Herpes Zoster vaccine (GSK1437173A)

INTERVENTIONS:
Biological: Herpes Zoster vaccine (GSK1437173A) — 2 doses administered intramuscularly in deltoid region of non-dominant arm.
  Other Names: HZ/su vaccine

SUMMARY:
The purpose of this study is to evaluate the immunogenicity and safety of GSK Biologicals' HZ/su vaccine in subjects' ≥ 50 years of age (YOA) who previously have had Herpes Zoster (HZ). The data collected will be compared with the data from subjects without HZ in other HZ/su trials.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a physician-documented history of HZ.
* Subjects who, in the opinion of the investigator, can and will comply with the requirements of the protocol.
* A male or female aged 50 years or older at the time of the first vaccination.
* Written informed consent obtained from the subject.
* Female subjects of non-childbearing potential may be enrolled in the study.

  * Non-childbearing potential is defined as pre-menarche, current tubal ligation, hysterectomy, ovariectomy or post-menopause.
* Female subjects of childbearing potential may be enrolled in the study, if the subject:

  * has practiced adequate contraception for 30 days prior to vaccination, and
  * has a negative pregnancy test on the day of vaccination, and
  * has agreed to continue adequate contraception during the entire treatment period and for 2 months after completion of the vaccination series.

Exclusion Criteria:

* Active Herpes Zoster infection (a case is considered no more active when all lesions have at least turned to crusts).
* Use of any investigational or non-registered product other than the study vaccine/product within 30 days preceding the first dose of study vaccine/product, or planned use during the study period.
* Chronic administration (defined as > 14 consecutive days) of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose. For corticosteroids, a prednisone dose of <20 mg/day, or equivalent, is allowed. Inhaled, topical and intra-articular corticosteroids are allowed.
* Administration of long-acting immune-modifying drugs within six months prior to the first vaccine dose or expected administration at any time during the study period.
* Administration or planned administration of a live vaccine in the period starting 30 days before the first dose of study vaccine and ending 30 days after the last dose of study vaccine, or, administration or planned administration of a non-replicating vaccine within 8 days prior to or within 14 days after either dose of study vaccine.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational vaccine/product.
* Previous vaccination against VZV or HZ and/or planned administration during the study of an HZ vaccine other than the study vaccine.
* Any confirmed or suspected immunosuppressive or immunodeficient condition resulting from disease or immunosuppressive/cytotoxic therapy.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccine/product.
* Acute disease and/or fever at the time of enrolment.

  * Fever is defined as temperature ≥ 37.5°C /99.5°F for oral, axillary or tympanic route, or ≥ 38.0°C /100.4°F on rectal route. The preferred route for recording temperature in this study will be oral.
  * Subjects with a minor illness (such as mild diarrhoea, mild upper respiratory infection) without fever may, be enrolled at the discretion of the investigator.
* Administration of immunoglobulins and/or any blood products within the 3 months preceding the first dose of study vaccine or planned administration during the study period.
* Any condition which, in the judgment of the investigator, would make intramuscular injection unsafe.
* Pregnant or lactating female.
* Female planning to become pregnant or planning to discontinue contraceptive precautions before Month 4 (i.e. 2 months after the last dose of study vaccine).

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2013-06-10; Primary Completion 2014-02-10 (Actual); Study Completion 2014-11-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (4):
- Canada (2):
  - GSK Investigational Site, Coquitlam, British Columbia
  - GSK Investigational Site, Pointe-Claire, Quebec
- Russia (2):
  - GSK Investigational Site, Barnaul
  - GSK Investigational Site, Yekaterinburg

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Godeaux O, Kovac M, Shu D, Grupping K, Campora L, Douha M, Heineman TC, Lal H. Immunogenicity and safety of an adjuvanted herpes zoster subunit candidate vaccine in adults >/= 50 years of age with a prior history of herpes zoster: A phase III, non-randomized, open-label clinical trial. Hum Vaccin Immunother. 2017 May 4;13(5):1051-1058. doi: 10.1080/21645515.2016.1265715. Epub 2017 Jan 9. PMID 28068212
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 116796 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 116796 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 116796 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 116796 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 116796 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 116796 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 116796 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Groups:
- GSK1437173A Group: Subjects who received GSK1437173A vaccine according to a 0, 2-month schedule, administered intramuscularly into the deltoid muscle of the non-dominant arm.
Period: Overall Study
Arm/Group | GSK1437173A Group
Started | 96
Completed | 93
Not Completed | 3
Not completed — Adverse Event | 1
Not completed — Consent Withdrawal | 2

BASELINE CHARACTERISTICS:
Arm/Group | GSK1437173A Group
Number analyzed (Participants) | 96
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.9 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63
  Male | 33
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White - Caucasian/European | 92
  Asian - Central/South Asian | 2
  Asian - Japanese | 1
  White - Arabic /North African | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Vaccine Responders for Anti-gE Antibodies as Determined by ELISA
Description: Vaccine response was defined as:
  For initially seronegative subjects, antibody concentration at post-vaccination ≥ 4 fold the cut-off for anti-gE [4x97 milli-international units per milliliter (mIU/mL)]; For initially seropositive subjects, antibody concentration at post-vaccination ≥ 4 fold the pre-vaccination antibody concentration.
Time Frame: At Month 3
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity, which included all evaluable subjects for whom data concerning immunogenicity outcome variables were available.
Measure: Count of Participants; unit: Participants
Groups:
- GSK1437173A Group: Subjects who received GSK1437173A vaccine according to a 0, 2-month schedule, administered intramuscularly (IM) in the deltoid of the non-dominant arm.
- GSK1437173A Group 50-59 YOA: Subgroup of subjects between 50 and 59 Years of Age (YOA) who received GSK1437173A vaccine according to a 0, 2-month schedule, administered intramuscularly (IM) in the deltoid of the non-dominant arm.
- GSK1437173A Group 60-69 YOA: Subgroup of subjects between 60 and 69 Years of Age (YOA) who received GSK1437173A vaccine according to a 0, 2-month schedule, administered intramuscularly (IM) in the deltoid of the non-dominant arm.
- GSK1437173A Group >=70 YOA: Subgroup of subjects of or above 70 Years of Age (YOA) who received GSK1437173A vaccine according to a 0, 2-month schedule, administered intramuscularly (IM) in the deltoid of the non-dominant arm.
Arm/Group | GSK1437173A Group | GSK1437173A Group 50-59 YOA | GSK1437173A Group 60-69 YOA | GSK1437173A Group >=70 YOA
Number analyzed (Participants) | 82 | 29 | 28 | 25
Participants | 74 | 26 | 26 | 22

2. Primary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = pain that prevented normal activity. Grade 3 redness/swelling = redness/swelling spreading beyond 100 millimeters (mm) of injection site.
Time Frame: Within 7 days (Day 0-6) after each vaccine dose and across doses
Population: The analysis was performed on the Total Vaccinated cohort, which included all subjects with at least one study vaccine administered and with the symptoms sheet filled in.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A Group
Number analyzed (Participants) | 95
Participants
  Any Pain, Dose 1: number analyzed (Participants) | 94
  Any Pain, Dose 1 | 61
  Grade 3 Pain, Dose 1: number analyzed (Participants) | 94
  Grade 3 Pain, Dose 1 | 3
  Any Redness, Dose 1: number analyzed (Participants) | 94
  Any Redness, Dose 1 | 17
  Grade 3 Redness, Dose 1: number analyzed (Participants) | 94
  Grade 3 Redness, Dose 1 | 0
  Any Swelling, Dose 1: number analyzed (Participants) | 94
  Any Swelling, Dose 1 | 12
  Grade 3 Swelling, Dose 1: number analyzed (Participants) | 94
  Grade 3 Swelling, Dose 1 | 0
  Any Pain, Dose 2: number analyzed (Participants) | 86
  Any Pain, Dose 2 | 56
  Grade 3 Pain, Dose 2: number analyzed (Participants) | 86
  Grade 3 Pain, Dose 2 | 5
  Any Redness, Dose 2: number analyzed (Participants) | 86
  Any Redness, Dose 2 | 22
  Grade 3 Redness, Dose 2: number analyzed (Participants) | 86
  Grade 3 Redness, Dose 2 | 2
  Any Swelling, Dose 2: number analyzed (Participants) | 86
  Any Swelling, Dose 2 | 13
  Grade 3 Swelling, Dose 2: number analyzed (Participants) | 86
  Grade 3 Swelling, Dose 2 | 0
  Any Pain, Across Doses | 70
  Grade 3 Pain, Across Doses | 8
  Any Redness, Across Doses | 31
  Grade 3 Redness, Across Doses | 2
  Any Swelling, Across Doses | 19
  Grade 3 Swelling, Across Doses | 0

3. Primary Outcome: Number of Days With Solicited Local Symptoms
Description: The number of days with any local symptoms during the solicited post-vaccination period.
Time Frame: Within 7 days (Day 0-6) after each vaccine dose
Population: The analysis was performed on the Total Vaccinated cohort, which included all subjects with at least one study vaccine administered and with results available for this assessment.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | GSK1437173A Group
Number analyzed (Participants) | 96
Days
  Pain post-Dose 1 | 3.0 [2.0 to 4.0]
  Pain post-Dose 2 | 3.0 [2.0 to 4.0]
  Redness post-Dose 1 | 3.0 [1.0 to 4.0]
  Redness post-Dose 2 | 2.5 [2.0 to 4.0]
  Swelling post-Dose 1 | 3.0 [1.5 to 4.5]
  Swelling post-Dose 2 | 2.0 [2.0 to 3.0]

4. Primary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were fatigue, gastrointestinal (nausea, vomiting, diarrhoea and/or abdominal pain), headache, myalgia, shivering and temperature [defined as oral temperature equal to or above 37.5 degrees Celsius (°C)]. Any = occurrence of the symptom regardless of intensity grade. Grade 3 symptom = symptom that prevented normal activity. Grade 3 temperature = temperature > 39.0 °C. Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: Within 7 days (Day 0-6) after each vaccine dose and across doses
Population: The analysis was performed on the Total Vaccinated cohort, which included all subjects with at least one dose of the study vaccine administered and with the symptoms sheet filled in.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A Group
Number analyzed (Participants) | 95
Participants
  Any Fatigue, Dose 1: number analyzed (Participants) | 94
  Any Fatigue, Dose 1 | 37
  Related Fatigue, Dose 1: number analyzed (Participants) | 94
  Related Fatigue, Dose 1 | 29
  Grade 3 Fatigue, Dose 1: number analyzed (Participants) | 94
  Grade 3 Fatigue, Dose 1 | 5
  Any Gastrointestinal, Dose 1: number analyzed (Participants) | 94
  Any Gastrointestinal, Dose 1 | 14
  Related Gastrointestinal, Dose 1: number analyzed (Participants) | 94
  Related Gastrointestinal, Dose 1 | 6
  Grade 3 Gastrointestinal, Dose 1: number analyzed (Participants) | 94
  Grade 3 Gastrointestinal, Dose 1 | 1
  Any Headache, Dose 1: number analyzed (Participants) | 94
  Any Headache, Dose 1 | 22
  Related Headache, Dose 1: number analyzed (Participants) | 94
  Related Headache, Dose 1 | 15
  Grade 3 Headache, Dose 1: number analyzed (Participants) | 94
  Grade 3 Headache, Dose 1 | 1
  Any Myalgia, Dose 1: number analyzed (Participants) | 94
  Any Myalgia, Dose 1 | 25
  Related Myalgia, Dose 1: number analyzed (Participants) | 94
  Related Myalgia, Dose 1 | 21
  Grade 3 Myalgia, Dose 1: number analyzed (Participants) | 94
  Grade 3 Myalgia, Dose 1 | 5
  Any Shivering, Dose 1: number analyzed (Participants) | 94
  Any Shivering, Dose 1 | 15
  Related Shivering, Dose 1: number analyzed (Participants) | 94
  Related Shivering, Dose 1 | 14
  Grade 3 Shivering, Dose 1: number analyzed (Participants) | 94
  Grade 3 Shivering, Dose 1 | 2
  Any Temperature/(Oral), Dose 1: number analyzed (Participants) | 94
  Any Temperature/(Oral), Dose 1 | 7
  Related Temperature/(Oral), Dose 1: number analyzed (Participants) | 94
  Related Temperature/(Oral), Dose 1 | 6
  Grade 3 Temperature/(Oral), Dose 1: number analyzed (Participants) | 94
  Grade 3 Temperature/(Oral), Dose 1 | 0
  Any Fatigue, Dose 2: number analyzed (Participants) | 86
  Any Fatigue, Dose 2 | 41
  Related Fatigue, Dose 2: number analyzed (Participants) | 86
  Related Fatigue, Dose 2 | 28
  Grade 3 Fatigue, Dose 2: number analyzed (Participants) | 86
  Grade 3 Fatigue, Dose 2 | 6
  Any Gastrointestinal, Dose 2: number analyzed (Participants) | 86
  Any Gastrointestinal, Dose 2 | 13
  Related Gastrointestinal, Dose 2: number analyzed (Participants) | 86
  Related Gastrointestinal, Dose 2 | 6
  Grade 3 Gastrointestinal, Dose 2: number analyzed (Participants) | 86
  Grade 3 Gastrointestinal, Dose 2 | 2
  Any Headache, Dose 2: number analyzed (Participants) | 86
  Any Headache, Dose 2 | 29
  Related Headache, Dose 2: number analyzed (Participants) | 86
  Related Headache, Dose 2 | 20
  Grade 3 Headache, Dose 2: number analyzed (Participants) | 86
  Grade 3 Headache, Dose 2 | 3
  Any Myalgia, Dose 2: number analyzed (Participants) | 86
  Any Myalgia, Dose 2 | 27
  Related Myalgia, Dose 2: number analyzed (Participants) | 86
  Related Myalgia, Dose 2 | 23
  Grade 3 Myalgia, Dose 2: number analyzed (Participants) | 86
  Grade 3 Myalgia, Dose 2 | 2
  Any Shivering, Dose 2: number analyzed (Participants) | 86
  Any Shivering, Dose 2 | 25
  Related Shivering, Dose 2: number analyzed (Participants) | 86
  Related Shivering, Dose 2 | 21
  Grade 3 Shivering, Dose 2: number analyzed (Participants) | 86
  Grade 3 Shivering, Dose 2 | 5
  Any Temperature/(Oral), Dose 2: number analyzed (Participants) | 86
  Any Temperature/(Oral), Dose 2 | 14
  Related Temperature/(Oral), Dose 2: number analyzed (Participants) | 86
  Related Temperature/(Oral), Dose 2 | 11
  Grade 3 Temperature/(Oral), Dose 2: number analyzed (Participants) | 86
  Grade 3 Temperature/(Oral), Dose 2 | 0
  Any Fatigue, Across Doses | 57
  Related Fatigue, Across Doses | 43
  Grade 3 Fatigue, Across Doses | 10
  Any Gastrointestinal, Across Doses | 23
  Related Gastrointestinal, Across Doses | 11
  Grade 3 Gastrointestinal, Across Doses | 2
  Any Headache, Across Doses | 37
  Related Headache, Across Doses | 28
  Grade 3 Headache, Across Doses | 4
  Any Myalgia, Across Doses | 35
  Related Myalgia, Across Doses | 31
  Grade 3 Myalgia, Across Doses | 6
  Any Shivering, Across Doses | 31
  Related Shivering, Across Doses | 26
  Grade 3 Shivering, Across Doses | 7
  Any Temperature/(Oral), Across Doses | 19
  Related Temperature/(Oral), Across Doses | 15
  Grade 3 Temperature/(Oral), Across Doses | 0

5. Primary Outcome: Number of Days With Solicited General Symptoms
Description: The number of days with general symptoms during the solicited post-vaccination period.
Time Frame: Within 7 days (Day 0-6) after each vaccine dose
Population: The analysis was performed on the Total Vaccinated cohort, which included all subjects with at least one dose of the study vaccine administered and with results available for this assessment.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | GSK1437173A Group
Number analyzed (Participants) | 96
Days
  Fatigue post-Dose 1 | 2.0 [1.0 to 4.0]
  Fatigue post-Dose 2 | 2.0 [1.0 to 3.0]
  Gastrointestinal symptoms post-Dose 1 | 1.5 [1.0 to 3.0]
  Gastrointestinal symptoms post-Dose 2 | 1.0 [1.0 to 2.0]
  Headache post-Dose 1 | 2.0 [1.0 to 3.0]
  Headache post-Dose 2 | 2.0 [1.0 to 3.0]
  Myalgia post-Dose 1 | 3.0 [2.0 to 4.0]
  Myalgia post-Dose 2 | 2.0 [1.0 to 3.0]
  Shivering post-Dose 1 | 1.0 [1.0 to 2.0]
  Shivering post-Dose 2 | 1.0 [1.0 to 2.0]
  Temperature post-Dose 1 | 1.0 [1.0 to 1.0]
  Temperature post-Dose 2 | 1.5 [1.0 to 2.0]

6. Primary Outcome: Number of Subjects With Any, Grade 3 and Related Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination. Grade 3 AE = an AE which prevented normal, everyday activities. Related = AE assessed by the investigator as related to the vaccination.
Time Frame: Within 30 days (Days 0-29) after each vaccination
Population: The analysis was performed on the Total Vaccinated cohort, which included all subjects with at least one dose of the study vaccine administered.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A Group
Number analyzed (Participants) | 96
Participants
  Any AE(s) | 30
  Grade 3 AE(s) | 11
  Related AE(s) | 12

7. Primary Outcome: Number of Subjects With Any Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life-threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: From first vaccination up to 30 days post last vaccination
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A Group
Number analyzed (Participants) | 96
Participants | 1

8. Primary Outcome: Number of Subjects With Any Potential Immune-mediated Diseases (pIMDs)
Description: Potential immune-mediated diseases (pIMDs) are a subset of AEs that include autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have an autoimmune aetiology.
Time Frame: From first vaccination up to 30 days post last vaccination
Population: The analysis was performed on the Total Vaccinated cohort, which included all subjects with at least one study vaccine administered.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A Group
Number analyzed (Participants) | 96
Participants | 0

9. Secondary Outcome: Anti-gE Antibody Concentrations
Description: Anti-gE antibody concentrations were presented as geometric mean concentrations (GMCs) and expressed in milli-international units per milliliter (mIU/mL). The outcome was assessed in each of the following age ranges: 50-59 YOA, 60-69 YOA and ≥ 70 YOA, in terms of antibody concentrations.
Time Frame: At Month 0 and at Month 3
Population: The analysis was performed on the ATP cohort for immunogenicity, which included all evaluable subjects for whom data concerning immunogenicity outcome variables were available.
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | GSK1437173A Group 50-59 YOA | GSK1437173A Group 60-69 YOA | GSK1437173A Group >=70 YOA
Number analyzed (Participants) | 29 | 28 | 25
mIU/mL
  Anti-gE at Month 0 | 2561.4 [1531.4 to 4284.2] | 2083.5 [1357.4 to 3198.0] | 2600.6 [1319.4 to 5125.9]
  Anti-gE at Month 3 | 56413.7 [43783.3 to 72687.6] | 44470.8 [37373.2 to 52916.2] | 42642.5 [34698.8 to 52404.9]

10. Secondary Outcome: Number of Subjects With Anti-gE Antibody Concentrations Equal to or Above the Cut-off Value
Description: The cut-off value was 97 mIU/mL.
Time Frame: At Month 0 and at Month 3
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A Group 50-59 YOA | GSK1437173A Group 60-69 YOA | GSK1437173A Group >=70 YOA
Number analyzed (Participants) | 29 | 28 | 25
Participants
  Anti-gE at Month 0 | 29 | 28 | 25
  Anti-gE at Month 3 | 29 | 28 | 25

11. Secondary Outcome: Number of Subjects With SAEs
Description: as for outcome 7
Time Frame: Starting after 30 days post last vaccination until study end (i.e. Month 14)
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A Group
Number analyzed (Participants) | 96
Participants | 2

12. Secondary Outcome: Number of Subjects With Any Potential Immune-mediated Diseases (pIMDs)
Description: as for outcome 8
Time Frame: Starting after 30 days post last vaccination until study end (i.e. Month 14)
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A Group
Number analyzed (Participants) | 96
Participants | 0

ADVERSE EVENTS:
Time Frame: Serious Adverse Events were assessed throughout the study (up to Month 14). Other Adverse Events were assessed during the 30-day (Days 0-29) post-vaccination period.
Arm/Group | GSK1437173A Group
All-Cause Mortality (participants affected / at risk) | 0/96
Serious Adverse Events (participants affected / at risk) | 3/96
Other Adverse Events (participants affected / at risk) | 77/96
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK1437173A Group (N=96)
Chronic gastritis (Gastrointestinal disorders) | 1 (1)
Duodenal ulcer perforation (Gastrointestinal disorders) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK1437173A Group (N=96)
Chills (General disorders) | 31 (42)
Erythema (Skin and subcutaneous tissue disorders) | 31 (39)
Fatigue (General disorders) | 57 (78)
Gastrointestinal disorder (Gastrointestinal disorders) | 23 (27)
Headache (Nervous system disorders) | 37 (51)
Myalgia (Musculoskeletal and connective tissue disorders) | 35 (52)
Pain (General disorders) | 70 (118)
Pyrexia (General disorders) | 19 (21)
Swelling (General disorders) | 19 (25)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.